CLINICAL TRIAL: NCT05311618
Title: A Phase 1/1b Dose Escalation/Expansion Study of NGM438 as Monotherapy and in Combination With Pembrolizumab in Advanced or Metastatic Solid Tumors
Brief Title: Study of NGM438 as Monotherapy and in Combination With Pembrolizumab in Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 438-IO-101; KEYNOTE-E20 (Other: Merck Sharp & Dohme LLC); MK-3475-E20 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2022-03-18; First posted 2022-04-05 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer; Breast Cancer; Gastric Cancer; Non Small Cell Lung Cancer; Cervical Cancer; Endocervical Cancer; Squamous Cell Carcinoma of Head and Neck; Bladder Urothelial Cancer; Colorectal Cancer; Esophageal Cancer; Ovarian Cancer; Renal Cell Carcinoma; Prostate Cancer; Melanoma; Mesothelioma; Cholangiocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Breast Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Esophageal Neoplasms; Ovarian Neoplasms; Carcinoma, Renal Cell; Prostatic Neoplasms; Melanoma; Mesothelioma; Cholangiocarcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NGM438 Monotherapy Dose Escalation (Experimental): Part 1a Single Agent Dose Escalation
  Interventions: Drug: NGM438
- NGM438 Combination Dose Finding with pembrolizumab ( KEYTRUDA ® ) (Experimental): Part 1b NGM438 plus pembrolizumab ( KEYTRUDA ® )
  Interventions: Drug: NGM438; Drug: Pembrolizumab (KEYTRUDA ®)
- Biopsy Cohort with NGM438 Monotherapy Followed by Combination Therapy with Pembrolizumab(KEYTRUDA ®) (Experimental): Part 1C NGM438 followed by NGM438 plus pembrolizumab ( KEYTRUDA ® )
  Interventions: Drug: NGM438; Drug: Pembrolizumab (KEYTRUDA ®)

INTERVENTIONS:
Drug: NGM438 — NGM438 is given intravenously (IV) every 3 weeks in a 21 day cycle. Multiple dose levels will be evaluated.
Drug: Pembrolizumab (KEYTRUDA ®) — Pembrolizumab (KEYTRUDA®) will be administered intravenously (IV) every 3 weeks in a 21 day cycle.
  Arms: Biopsy Cohort with NGM438 Monotherapy Followed by Combination Therapy with Pembrolizumab(KEYTRUDA ®); NGM438 Combination Dose Finding with pembrolizumab ( KEYTRUDA ® )

SUMMARY:
Study of NGM438 as Monotherapy and in Combination with Pembrolizumab in Advanced or Metastatic Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced or metastatic solid tumor malignancy.
* Progressed or was intolerant to all available therapies known to confer clinical benefit appropriate for their tumor type for which the patient was eligible and willing to receive.
* Adequate bone marrow, kidney and liver function
* Performance status of 0 or 1.
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade 1 except for AEs not constituting a safety risk by Investigator judgement.

Exclusion Criteria:

• Prior treatment targeting LAIR1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose-limiting Toxicities | Baseline up to 21 Days
  A DLT is defined as an AE that meets at least one of the criteria listed in protocol, according to National Cancer Institute (NCI) common terminology criteria for AE (CTCAE) version 5.0, and is considered by the Investigator to be clinically relevant and attributed to the study treatment during the first 21 days after the first dose of study treatment.
Number of Patients with Adverse Events | Approximately 24 months
  Number of patients with adverse events (AEs) according to severity, seriousness, and relationship to study drug.
  An AE is defined as any untoward medical occurrence in a patient, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of patients who experience at least one AE will be presented.
Number of Patients with Clinically Significant Laboratory Abnormalities | Approximately 24 months
  Number of patients with clinically significant change from baseline in laboratory abnormalities as characterized by type, frequency, severity (graded by CTCAE version 5.0) and timing.
Changes in potential pharmacodynamic biomarker CD163 in paired tumor tissue in Patients in the Biopsy Cohort Summary of baseline, post baseline and changes from baseline in CD163 | Baseline up to 15 days
Changes in potential pharmacodynamic biomarker MMP9 in paired tumor tissue in Patients in the Biopsy Cohort Summary of baseline, post baseline and changes from baseline in MMP9 | Baseline up to 15 days
Changes in potential pharmacodynamic biomarker CD8 in paired tumor tissue in Patients in the Biopsy Cohort Summary of baseline, post baseline and changes from baseline in CD8 | Baseline up to 15 days

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of NGM438 | Approximately 24 months. Each Cycle is 21 days.
  Cmax is defined as the observed maximum serum concentration post drug administration.
  Will be measured on Day 1, 2, 4, 8 and 15 of Cycles 1 and 3, Day 1 of Cycle 2 and Day 1 of Cycles 4-6 and every third cycle thereafter
Area Under the Curve (AUC) of Serum NGM438 | Approximately 24 months. Each Cycle is 21 days.
  Area under the curve from time zero extrapolated to the last time point prior to the next dose.
  Will be measured on Day 1, 2, 4, 8 and 15 of Cycles 1 and 3, Day 1 of Cycle 2 and Day 1 of Cycles 4-6 and every third cycle thereafter
Time to Maximum (Tmax) Observed Serum Concentration of NGM438 | Approximately 24 months. Each Cycle is 21 days.
  Tmax is defined as the time to reach the observed maximum serum concentration (Cmax).
  Will be measured on Day 1, 2, 4, 8 and 15 of Cycles 1 and 3, Day 1 of Cycle 2 and Day 1 of Cycles 4-6 and every third cycle thereafter
Half-life (t1/2) of NGM438 in Serum | Approximately 24 months. Each Cycle is 21 days.
  Time measured for the serum concentration to decrease by one half during the terminal phase.
  Will be measured on Day 1, 2, 4, 8 and 15 of Cycles 1 and 3, Day 1 of Cycle 2 and Day 1 of Cycles 4-6 and every third cycle thereafter
Systemic Clearance (CL) of NGM438 | Approximately 24 months. Each Cycle is 21 days.
  CL is defined as systemic clearance. Will be measured on Day 1, 2, 4, 8 and 15 of Cycles 1 and 3, Day 1 of Cycle 2 and Day 1 of Cycles 4-6 and every third cycle thereafter
Volume of Distribution (Vss) of NGM438 at Steady State | Approximately 24 months. Each Cycle is 21 days.
  Vss is defined as the volume of distribution at steady state. Will be measured on Day 1, 2, 4, 8 and 15 of Cycles 1 and 3, Day 1 of Cycle 2 and Day 1 of Cycles 4-6 and every third cycle thereafter
Anti-drug Antibodies (ADA) Against NGM438 | Approximately 24 months. Each Cycle is 21 days.
  Incidence and titers of anti-drug antibodies (ADA) against NGM438. Will be measured on Day 1 of each cycle through Cycle 6 and every third cycle thereafter.
Number of Patients in Dose Escalation and Dose Finding Cohorts with Objective Responses | Approximately 24 months
  Objective Response Rate is defined as the proportion of patients who achieve a confirmed complete response (CR) or partial response (PR) divided by the total number of evaluable patients per RECIST v1.1
Trough Concentrations of NGM438 in Patients in the Biopsy Cohort | Approximately 24 months. Each Cycle is 21 days.
  Trough Concentration refers to the serum concentration of NGM438 observed just before treatment administration.
  Will be measured on Day 1, 2, 4, 8 and 15 of Cycles 1 and 3, Day 1 of Cycle 2 and Day 1 of Cycle 4 and each cycle thereafter.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - SCRI Denver, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Henry Ford Health System, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Mount Sinai Hospital, New York, New York
  - MD Anderson, Houston, Texas